CLINICAL TRIAL: NCT04317066
Title: A Phase 1 Clinical Study of Pembrolizumab (MK-3475) in Participants With Relapsed or Refractory Primary Mediastinal Large B-cell Lymphoma (rrPMBCL) (KEYNOTE-A33)
Brief Title: A Study of Pembrolizumab (MK-3475) in Participants With Relapsed or Refractory Primary Mediastinal Large B-cell Lymphoma (rrPMBCL) (MK-3475-A33/KEYNOTE-A33)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 3475-A33; MK-3475-A33 (Other: MSD); KEYNOTE-A33 (Other: MSD); 205262 (Registry Identifier: Japic-CTI); 2080225167 (Other: JRCT)
Record Dates: First submitted 2020-03-19; First posted 2020-03-20 (Actual); Results first posted 2025-04-06 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-03

CONDITIONS: Lymphoma, B-Cell
Keywords: Programmed Cell Death-1 (PD1, PD-1); Programmed Death-Ligand 1 (PDL1, PD-L1)
MeSH Terms: conditions — Lymphoma, B-Cell; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab in Participants with rrPMBCL (Experimental): Participants with relapsed or refractory primary mediastinal large B-cell lymphoma (rrPMBCL) receive Pembrolizumab 200 mg by intravenous (IV) infusion on day 1 of each 3-week cycle for up to 35 cycles (approximately 2 years).
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab 200 mg by intravenous (IV) infusion, given on day 1 of each 3-week cycle.
  Other Names: KEYTRUDA®; MK-3475

SUMMARY:
The purpose of this study is to evaluate the objective response, safety, and tolerability of pembrolizumab in Japanese participants who have refractory primary mediastinal large B-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Primary mediastinal B-cell lymphoma (PMBCL)
* Relapsed or refractory PMBCL and:

  * Relapsed after auto-stem cell transplantation (SCT) or have failed to achieve a complete response (CR) or partial response (PR) within 60 days of auto-SCT; or
  * For participants who are ineligible for auto-SCT, has received at least ≥ 2 lines of prior therapy and have failed to respond to or relapsed after their last line of treatment. For participants who received consolidative local radiotherapy after systemic therapy, local radiotherapy will not be considered as a separate line of treatment
* Previously exposed to rituximab as part of prior lines of treatment
* Radiographically measurable disease
* Performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale
* Life expectancy ≥3 months
* Adequate organ function
* Male participants of childbearing potential must agree to use an adequate method of contraception, starting with the first dose of study drug through 120 days after the last dose of study drug, OR must be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent
* Female participants of childbearing potential must be willing to use an adequate method of contraception for the course of the study through 120 days after the last dose of study drug OR must be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent

Exclusion Criteria:

* Received prior therapy with an anti-PD-1 (programmed cell death protein 1), anti-PD-L1 (programmed death-ligand 1), or anti-PD-L2 (programmed cell death 1 ligand 2), or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4 [cytotoxic T-lymphocyte-associated protein 4], OX 40, or CD137 [cluster of differentiation 137])
* Received chimeric antigen receptor (CAR) T-cell therapy
* Prior monoclonal antibody or radiation therapy within 4 weeks prior to the first dose of study intervention; OR received prior chemotherapy or targeted small molecule therapy within 2 weeks prior to the first dose of study intervention; OR has not recovered from adverse events due to a previously administered agent above. Participants with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study
* Major surgery within 3 weeks prior to first dose of study intervention
* Received a live vaccine within 30 days prior to the first dose of study drug
* Currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study intervention Participants in the follow-up phase of an investigational study may participate as long as it has been 4 weeks after the last dose of the previous investigational agent
* Diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior the first dose of study drug
* Known additional malignancy that is progressing or has required active treatment within the past 3 years. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or carcinoma in situ, that have undergone potentially curative therapy
* Known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients
* Active autoimmune disease that has required systemic treatment in past 2 years
* History of (non-infectious) pneumonitis that required steroids, or current pneumonitis
* Active infection requiring systemic therapy
* History of human immunodeficiency virus (HIV) or Hepatitis B
* Active Hepatitis C virus infection
* Known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study
* Pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study intervention
* Allogeneic hematopoietic stem cell/solid organ transplantation within the last 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2020-06-26 (Actual); Primary Completion 2024-04-11 (Actual); Study Completion 2024-04-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (9):
- Japan (9):
  - Nagoya University Hospital ( Site 0002), Nagoya, Aichi-ken
  - Hokkaido University Hospital ( Site 0006), Sapporo, Hokkaido
  - Kindai University Hospital ( Site 0001), Sayama, Osaka
  - National Hospital Organization Disaster Medical Center ( Site 0007), Tachikawa, Tokyo
  - Kyushu University Hospital ( Site 0008), Fukuoka
  - Okayama University Hospital ( Site 0004), Okayama
  - National Cancer Center Hospital ( Site 0005), Tokyo
  - Tokyo Metropolitan Komagome Hospital ( Site 0009), Tokyo
  - Yamagata University Hospital ( Site 0003), Yamagata

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Kato K, Nakamura S, Wakana A, Koh Y, Izutsu K. Pembrolizumab in Japanese patients with primary mediastinal large B-cell lymphoma: results from the KEYNOTE-A33 study. Int J Clin Oncol. 2024 Dec;29(12):1977-1983. doi: 10.1007/s10147-024-02627-8. Epub 2024 Sep 18. PMID 39294486
- See also: Merck Clinical Trials Information — https://merckclinicaltrials.com/

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All allocated participants.
Groups:
- Pembrolizumab in Participants With rrPMBCL: Participants with relapsed or refractory primary mediastinal large B-cell lymphoma (rrPMBCL) received Pembrolizumab 200 mg by Intravenous (IV) infusion on day 1 of each 3-week cycle for up to 35 cycles (approximately 2 years).
Period: Overall Study
Arm/Group | Pembrolizumab in Participants With rrPMBCL
Started | 7
Completed | 0
Not Completed | 7
Not completed — Sponsor decision | 5
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Arm/Group | Pembrolizumab in Participants With rrPMBCL
Number analyzed (Participants) | 7
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.3 (6.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 7
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 7
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR) Using International Working Group (IWG) Revised Response Criteria for Malignant Lymphoma as Assessed by Independent Central Review
Description: ORR is defined as the percentage of participants with response (complete response, CR or partial response, PR) according to the International Working Group (IWG) Response Assessment Criteria for Malignant Lymphoma per Cheson 2007. CR is the disappearance of all evidence of disease. PR is ≥ 50% decrease in the sum of product diameters (SPD) of the six largest dominant nodes or nodal masses, ≥ 50% decrease in SPD of splenic and hepatic nodules, no increase in the size of the other nodes, liver, or spleen plus no measurable disease in other organs and no new sites of disease. Per protocol, the percentage of participants who experienced a CR or PR as assessed by independent central review were reported.
Time Frame: Up to approximately 24 months
Population: The analysis population consisted of all participants who received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab in Participants With rrPMBCL
Number analyzed (Participants) | 7
Percentage of Participants | 42.9 [9.9 to 81.6]

2. Primary Outcome: Number of Participants Who Experienced at Least One Adverse Event (AE)
Description: An adverse event (AE) was defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, which occurs during the course of the study. Per protocol, the number of participants who experienced at least one AE were reported.
Time Frame: Up to approximately 27 months
Population: The analysis population consisted of all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab in Participants With rrPMBCL
Number analyzed (Participants) | 7
Participants | 7

3. Primary Outcome: Number of Participants Who Discontinued Study Treatment Due to an Adverse Event (AE)
Description: An AE was defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, which occurs during the course of the study. Per protocol, the number of participants who discontinued study treatment due to an AE were reported.
Time Frame: Up to approximately 24 months
Population: The analysis population consisted of all participants who received at least 1 dose of study treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab in Participants With rrPMBCL
Number analyzed (Participants) | 7
Participants | 0

4. Secondary Outcome: Objective Response Rate (ORR) Using International Working Group (IWG) Revised Response Criteria for Malignant Lymphoma as Assessed by Investigator
Description: ORR is defined as the percentage of participants with response (complete response, CR or partial response, PR) according to the International Working Group (IWG) Response Assessment Criteria for Malignant Lymphoma per Cheson 2007. CR is the disappearance of all evidence of disease. PR is ≥ 50% decrease in the sum of product diameters (SPD) of the six largest dominant nodes or nodal masses, ≥ 50% decrease in SPD of splenic and hepatic nodules, no increase in the size of the other nodes, liver, or spleen plus no measurable disease in other organs and no new sites of disease. Per protocol, the percentage of participants who experienced a CR or PR as assessed by investigator review were reported.
Time Frame: Up to approximately 24 months
Population: The analysis population consisted of all participants who received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab in Participants With rrPMBCL
Number analyzed (Participants) | 7
Percentage of Participants | 57.1 [18.4 to 90.1]

5. Secondary Outcome: Disease Control Rate (DCR) Using International Working Group (IWG) Revised Response Criteria for Malignant Lymphoma as Assessed by Independent Central Review
Description: The DCR was defined as the percentage of participants in the analysis population who have achieved a CR, PR or stable disease (SD) response prior to PD according to the International Working Group (IWG) Response Assessment Criteria for Malignant Lymphoma per Cheson 2007. CR is the disappearance of all evidence of disease and PR is the regression of measurable disease and no new sites of disease. SD is the failure to attain CR/PR or PD. PD is the appearance any new lesion or increase by ≥ 50% of previously involved site from nadir. Per protocol, the percentage of participants who experienced a CR, a PR, or SD as assessed by independent central review were reported.
Time Frame: Up to approximately 24 months
Population: The analysis population consisted of all participants who received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab in Participants With rrPMBCL
Number analyzed (Participants) | 7
Percentage of Participants | 57.1 [18.4 to 90.1]

6. Secondary Outcome: Disease Control Rate (DCR) Using International Working Group (IWG) Revised Response Criteria for Malignant Lymphoma as Assessed by Investigator
Description: The DCR was defined as the percentage of participants in the analysis population who have achieved a CR, PR or stable disease (SD) response prior to PD according to the International Working Group (IWG) Response Assessment Criteria for Malignant Lymphoma per Cheson 2007. CR is the disappearance of all evidence of disease and PR is the regression of measurable disease and no new sites of disease. SD is the failure to attain CR/PR or PD. PD is the appearance any new lesion or increase by ≥ 50% of previously involved site from nadir. Per protocol, the percentage of participants who experienced a CR, a PR, or SD as assessed by investigator review were reported.
Time Frame: Up to approximately 24 months
Population: The analysis population consisted of all participants who received at least 1 dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Pembrolizumab in Participants With rrPMBCL
Number analyzed (Participants) | 7
Percentage of Participants | 71.4 [29 to 96.3]

ADVERSE EVENTS:
Time Frame: Up to approximately 27 months
Description: All-Cause Mortality, serious and non-serious adverse events (AEs) were reported on all allocated participants who received at least 1 dose of study treatment.
Arm/Group | Pembrolizumab in Participants With rrPMBCL
All-Cause Mortality (participants affected / at risk) | 2/7
Serious Adverse Events (participants affected / at risk) | 1/7
Other Adverse Events (participants affected / at risk) | 7/7
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab in Participants With rrPMBCL (N=7)
Adrenal insufficiency (Endocrine disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab in Participants With rrPMBCL (N=7)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Neutropenia (Blood and lymphatic system disorders) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (5)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Haemorrhoids (Gastrointestinal disorders) | 1 (1)
Malaise (General disorders) | 1 (1)
Pyrexia (General disorders) | 3 (3)
Hypersensitivity (Immune system disorders) | 1 (1)
Conjunctivitis (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 2 (2)
Paronychia (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Alanine aminotransferase increased (Investigations) | 2 (3)
Aspartate aminotransferase increased (Investigations) | 2 (3)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all manuscripts or abstracts before submission. Any information identified by the sponsor as confidential must be deleted prior to submission.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-11-28): https://cdn.clinicaltrials.gov/large-docs/66/NCT04317066/Prot_SAP_000.pdf